CLINICAL TRIAL: NCT03902613
Title: 18F-DOPA PET to Elucidate the Antidepressant Mechanism of Lurasidone in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Martin Lan, Assistant Professor of Psychiatry at CUMC, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7673
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lurasidone (Experimental): Open-label treatment with lurasidone within the dose range of 20-60 mg daily
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Participant will have an open label trial of lurasidone for eight weeks.

SUMMARY:
The goal of this project is to understand what causes bipolar disorder and how medications treat bipolar depression. Particularly, the project focuses on the importance of dopamine signaling in the process. Participants will have two different brain scans (MRI and PET scan). They will also have treatment for your depression with an FDA approved medication, lurasidone (Latuda). The study is funded by the Columbia University Irving Institute to improve the treatment of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I disorder, bipolar II disorder or other specified bipolar disorder
* Currently in a major depressive episode and moderately depressed
* Age 18-50 years old
* Patients on psychiatric medications will not be benefitting from those medications
* Females of childbearing potential must be willing to use an acceptable form of birth control throughout the study

Exclusion Criteria:

* Diagnosis of schizophrenia or other psychotic disorders, recent alcohol or substance use disorder, recent anorexia or bulimia nervosa
* Previous failed trial of lurasidone, or had intolerable side effects of lurasidone
* Significant active physical illness
* Actively suicidal
* ECT within the past 6 months
* Recent pregnancy, abortion or miscarriage or plans to conceive during the study; currently lactating
* Metal in the body that is not MRI compatible
* Current, past or anticipated exposure to radiation
* Currently taking an anticoagulant medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lan, MD PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 46 [46 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: Measures severity of depression symptoms; Scale from 0 to 54; higher numbers mean greater depression severity, so a decrease in score is a better outcome.
Time Frame: 15 minutes
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 1
units on a scale | 34 [34 to 34]

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Lurasidone
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03902613/Prot_SAP_000.pdf